CLINICAL TRIAL: NCT01499602
Title: LNG-IUS or Norethisterone Acetate for Treatment of Non-atypical Endometrial Hyperplasia in Perimenopausal Women
Brief Title: Efficacy of LNG-IUS for Treatment of Non-atypical Endometrial Hyperplasia in Perimenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hatem AbuHashim, Associate Professor of Obstetrics & Gynecology., Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-324v
Record Dates: First submitted 2011-12-20; First posted 2011-12-26 (Estimated); Last update posted 2011-12-26 (Estimated); Status verified 2011-12

CONDITIONS: Endometrial Hyperplasia
Keywords: Endometrial hyperplasia,; LNG-IUS,; Progestin
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — Levonorgestrel; Norethindrone Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LNG-IUS (Experimental): Release rate of 20µg Levonorgestrel(Mirena, Bayer Schering Pharma Oy, Finland) per day with one year follow up.
  Interventions: Drug: LNG-IUS; Mirena; Bayer Schering Pharma Oy, Finland
- Norethisterone Acetate (Active Comparator): Norethisterone Acetate tablets at a dose of 5 mg three times daily (15mg/day) for 3 weeks over three months.With persistence of endometrial hyperplasia, the treatment is repeated for another 3 months
  Interventions: Drug: Norethisterone Acetate tablets

INTERVENTIONS:
Drug: LNG-IUS; Mirena; Bayer Schering Pharma Oy, Finland — Initial release rate of 20µg Levonorgestrel per day for one year follow up.
  Arms: LNG-IUS
Drug: Norethisterone Acetate tablets — Norethisterone Acetate tablets at a dose of 5 mg three times daily (15mg/day) for 3 weeks over three months.With persistence of endometrial hyperplasia, the treatment is repeated for another 3 months
  Arms: Norethisterone Acetate

SUMMARY:
The purpose of this study is to compare the efficacy of the Levonorgestrel releasing Intrauterine System (Mirena) and Norethisterone Acetate for treatment of non-atypical endometrial hyperplasia in perimenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed simple or complex endometrial hyperplasia without atypia

Exclusion Criteria:

* Endometrial hyperplasia with atypia
* Other pathology e.g. patients with fibroids of any size, genital infection, adnexal abnormality.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2009-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in endometrial histopathology pattern from endometrial hyperplasia into regression status. | At 3 and 6 months

SECONDARY OUTCOMES:
Time to achieve complete regression | During the follow up period at 3,6,12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD. MRCOG, Principal Investigator — Mansoura University Hospital
Locations (1):
- Mansoura University Hospitals,OB/GYN department, Al Mansurah, Dakahlia Governorate, Egypt

REFERENCES:
- [Background] Reed SD, Voigt LF, Newton KM, Garcia RH, Allison HK, Epplein M, Jordan D, Swisher E, Weiss NS. Progestin therapy of complex endometrial hyperplasia with and without atypia. Obstet Gynecol. 2009 Mar;113(3):655-662. doi: 10.1097/AOG.0b013e318198a10a. PMID 19300331
- [Background] Lee SY, Kim MK, Park H, Yoon BS, Seong SJ, Kang JH, Jun HS, Park CT. The effectiveness of levonorgestrel releasing intrauterine system in the treatment of endometrial hyperplasia in Korean women. J Gynecol Oncol. 2010 Jun;21(2):102-5. doi: 10.3802/jgo.2010.21.2.102. Epub 2010 Jun 30. PMID 20613900